CLINICAL TRIAL: NCT06488989
Title: Left Bundle Branch Area Pacing in Patients With Heart Failure
Acronym: LBBAPHF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Center for Cardiac Surgery, Kazakhstan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol V1 (12.12.2023)
Record Dates: First submitted 2024-06-25; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Left Bundle Branch Area Pacing; Heart Failure; Cardiac Resynchronization Therapy; Cardiac Resynchronization Therapy Devices; Conduction System Pacing; Left Bundle-Branch Block
Keywords: heart failure; left bundle branch block; left bundle branch area pacing; medtronic; cardiac resynchronization therapy; kazakhstan
MeSH Terms: conditions — Heart Failure; Bundle-Branch Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with heart failure and left bundle branch block (Other): 1. Male or female ≥ 18 years of age at Visit 1.
  2. Patients with complete left bundle branch block, QRS duration greater than 130 ms, left ventricular ejection fraction (LVEF) less than 35%, and New York Heart Association (NYHA) functional class 2-3, who have been ineffective on optimal medical therapy for at least 3 months.
  3. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.
  Interventions: Device: left bundle branch area pacing

INTERVENTIONS:
Device: left bundle branch area pacing — Cardiac resynchronization therapy obtained by conduction system pacing

SUMMARY:
The relevance of Left Bundle Branch Pacing (LBBP) lies in its potential as a promising treatment option for patients with heart failure and left bundle branch block. LBBP aims to restore the normal physiological activation of the heart by delivering electrical impulses to the anatomical area of the left bundle branch, which may lead to more effective and synchronized ventricular contractions. Compared to traditional cardiac resynchronization therapy (CRT), this can result in a more physiological correction of dyssynchrony, improvement in left ventricular pump function, reduction in left ventricular volumes, and a decrease in mitral regurgitation. A crucial criterion is the reduction of heart failure symptoms and the enhancement of the patients quality of life.

DETAILED DESCRIPTION:
The aim The aim of Left Bundle Branch Pacing (LBBP) research is to assess its effectiveness in improving the contractile capacity of the left ventricular myocardium. The objectives are as follows

* To determine the optimal patient selection criteria;
* To assess long-term outcomes;
* To investigate safety and complications;
* To compare selective Left Bundle Branch Pacing (LBBP) with traditional cardiac resynchronization therapy in patients with heart failure.

Materials and Methods:

Materials: The study will include patients who were hospitalized at the National Research Cardiac Surgery Center (NRCS) in Astana, Kazakhstan. The study will be a mixed-methods approach, consisting of a retrospective component and a prospective component. The retrospective part of the study will involve the analysis of clinical and functional data of patients with left bundle branch block and heart failure. The prospective part of the study will involve the evaluation of quantitative and qualitative parameters based on transthoracic echocardiography data, the functional status of patients after LBBP implantation, and the assessment of long-term outcomes of the study, including its impact on mortality, hospitalization rates, and overall prognosis.

Inclusion Criteria:

* patients with complete left bundle branch block, QRS duration greater than 150 ms, left ventricular ejection fraction (LVEF) less than 35%, and New York Heart Association (NYHA) functional class 2-3, who have been ineffective on optimal medical therapy for at least 3 months.
* patients aged 18 years or older.
* Signed informed consent and willingness to collaborate with the researchers.

Exclusion Criteria:

- patient refusal to participate in the study.

Control Group:

patients post-implantation of traditional CRT-D.

Methods:

* Electrocardiography (ECG).
* Transthoracic echocardiography (EchoCG).
* 6-minute walk test.
* NT-proBNP measurement.
* Questionnaire-based assessments: SF-36, EQ-5D-5L.

Scientific Novelty:

This method is distinguished by its ability to provide highly physiological synchronized myocardial stimulation by stimulating the anatomical area of the left bundle branch, offering advantages such as shortening the ventricular electrical systole.

Advantages of the Method:

* Shortens ventricular electrical systole.
* Expands the possibilities of cardiac pacing in heart failure patients, including those who cannot undergo traditional cardiac resynchronization therapy (CRT) due to anatomical constraints (vascular anatomy) or other factors.
* LBBP can be considered as an alternative resynchronization method for non-responders to traditional CRT.

Practical Significance:

The procedure is simpler (less technically complex), electrode fixation is easier, the procedure duration and fluoroscopy time are shorter, it has the ability to maintain and improve left ventricular synchrony, and a shorter learning curve. Inclusion Criteria

1. Male or female ≥ 18 years of age at Visit 1.
2. patients with complete left bundle branch block, QRS duration greater than 130 ms, left ventricular ejection fraction (LVEF) less than 35%, and New York Heart Association (NYHA) functional class 2-3, who have been ineffective on optimal medical therapy for at least 3 months.
3. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.

Exclusion Criteria

1. Pregnancy.
2. Psychic disturbances.
3. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data - life expectancy less than 1 year.

Anticipated amount of patients - 50. STUDY TREATMENTS AND INTERVENTIONS day 1 - admission to cardiology department, acquisition of medical history, physical examination, blood tests, ECG, transthoracic echoCG.

day 2 - additional examinations (if necessary, depend on comorbidity), preparing for interventional procedure.

day 3 - implantation of cardiac resynchronization therapy device using Left bundle branch area pacing (LBBAP).

Procedure description:

LBBAP procedure was performed as previously described by Huang in 2017 and Ponnusamy in 2022. Monitoring of 12-lead ECG and intracardiac electrograms were performed utilizing WorkMate Claris electrophysiology system (Abbott, Plymouth, MN). DF-1 Implantable cardioverter-defibrillator (ICD) lead was placed into the right ventricle (RV) apex in all patients. LBBAP was performed using two types of leads and delivery catheters: C315HIS sheath with 3830 SelectSecure lead (Medtronic, Minneapolis, MN), and Selectra 3D with Solia S60 lead (Biotronik, Berlin, Germany). Left conduction system capture was confirmed in appliance with European Heart Rhythm Association (EHRA) clinical consensus statement on conduction system pacing implantation [10]. Main criteria to accept LBB area capture were: presence of terminal R-wave in lead V1; transition in QRS morphology from non-selective to selective during threshold test; short and stable V6 R-wave peak time (V6RWPT)<80 ms in different pacing outputs; V6-V1 interpeak>33 ms; sudden increase in V1 R-wave peak time (V1RWPT)>10 ms, split of EGM during threshold test.

day 4 - chest X-ray, device pocket ultrasound, device interrogation with lead testing, ECG.

day 5 - discharge from the hospital.

A Schedule of Events representing the required testing procedures to be performed for the duration of the study is diagrammed in Appendix 1.

Prior to conducting any study-related activities, written informed consent must be signed and dated by the subject or subject's legal representative. If appropriate, assent must also be obtained prior to conducting any study-related activities.

EVALUATIONS BY VISIT Visit 1 (admission to the hospital)

1. Review the study with the subject (subject's legal representative) and obtain written informed consent.
2. Assign the subject a unique screening number.
3. Record demographics data.
4. Record medical history, including a history of congestive heart failure, diagnosis date, and prior treatments.
5. Record concomitant medications.
6. Perform a complete physical examination.
7. Perform and record vital signs.
8. Perform and record oximetry.
9. Perform and record results of blood pressure testing.
10. Collect blood for clinical laboratory tests (chemistry, hematology, prothrombin time, NTPROBNP).
11. Obtain an echocardiogram, ECG.
12. Obtain a chest x-ray.
13. Implantation of device
14. Chest X-ray, ECG and device telemetry at 1 day after procedure
15. Discharge from the hospital and schedule subject for Visit 2 in 3 months. Visit 2 (3 months after discharge)

1. Record any Adverse Experiences and/or Review subject diary for adverse experiences 2. Perform abbreviated physical examination. 3. Perform and record vital signs. 4. Obtain an echocardiogram, ECG, chest X-ray. 5. NTproBNP test 6. ^ minute walk test (6MWT) 7. Questionnaire-based assessments: SF-36, EQ-5D-5L. 8. Device telemetry. Visit 3 (6 months after discharge)

1. Record any Adverse Experiences and/or Review subject diary for adverse experiences
2. Perform abbreviated physical examination.
3. Perform and record vital signs.
4. Obtain an echocardiogram, ECG, chest X-ray.
5. NTproBNP test
6. 6MWT
7. Questionnaire-based assessments: SF-36, EQ-5D-5L.
8. Device telemetry. Visit 4 (12 months after discharge)

1. Record any Adverse Experiences and/or Review subject diary for adverse experiences 2. Perform abbreviated physical examination. 3. Perform and record vital signs. 4. Obtain an echocardiogram, ECG, chest X-ray. 5. NTproBNP test 6. 6MWT 7. Questionnaire-based assessments: SF-36, EQ-5D-5L. 8. Device telemetry.

STATISTICAL METHODS AND CONSIDERATIONS This will be a non-randomized, prospective, single-centre, observational study. Participant characteristics and sequencing results will be summarized with descriptive statistics, including medians, averages, and standard deviations for continuous data. For categorical data, proportions with a 95% confidence interval will be calculated by the Klopper-Pearson method. Demographic, clinical and pathological characteristics will be compared using the criterion χ2 (categorical variables) and t-test/analysis of variance (continuous variables).Values of p<0.05 will be considered significant.

DATA COLLECTION, RETENTION AND MONITORING Data Collection Instruments The Investigator will prepare and maintain adequate and accurate source documents designed to record all observations and other pertinent data for each subject treated with the study drug.

Study personnel will enter data from source documents corresponding to a subject's visit into the protocol-specific electronic Case Report Form (eCRF) and paper CRF when the information corresponding to that visit is available. Subjects will not be identified by name in the study database but will be identified by a site number, subject number and initials.

For eCRFs: If a correction is required for an eCRF, the time and date stamps track the person entering or updating eCRF data and creates an electronic audit trail. For paper CRFs: If a correction is made on a CRF, the study staff member will line through the incorrect data, write in the correct data and initial and date the change.

The Investigator is responsible for all information collected on subjects enrolled in this study. All data collected during the course of this study must be reviewed and verified for completeness and accuracy by the Investigator. A copy of the CRF will remain at the Investigator's site at the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age at Visit 1.
2. Patients with complete left bundle branch block, QRS duration greater than 130 ms, left ventricular ejection fraction (LVEF) less than 35%, and New York Heart Association (NYHA) functional class 2-3, who have been ineffective on optimal medical therapy for at least 3 months.
3. Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

1. Pregnancy.
2. Psychic disturbances.
3. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data - life expectancy less than 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
General complications related to implantable cardiac device | From enrollment to the end of follow-up period at 12 months
  Incidence and amount of participants with general complication (deaths, stroke, thromboembolic complications);
procedure-related complications related to implantable cardiac device | From enrollment to the end of follow-up period at 12 months
  Incidence and amount of participants with procedure-related complication (pneumothorax, pocket/wound infection, systemic infection, pocket hematoma, atrial lead dislodgement, pericardial effusion, large vein thrombosis, re-intervention for other non-LBBAP lead reasons, subclavian arteriovenous fistula after puncture)
LBBAP lead-related complications complications related to implantable cardiac device | From enrollment to the end of follow-up period at 12 months
  Incidence and amount of patients with LBBAP lead-related complications (intraprocedural perforation into the left ventricle (LV) cavity , delayed perforation into the LV cavity, acute chest pain, acute ST-segment elevation in multiple leads, acute coronary syndrome, coronary vein fistula, coronary artery fistula, painful pacing/chest pain, right bundle branch injury, LBBAP lead unscrewable/trapped/damaged helix, LBBAP lead dislodgement, threshold rise to an absolute value > 2 V, threshold rise > 1 V from baseline, threshold rise leading to re-intervention)
shortening of QRS | From enrollment to the end of follow-up period at 12 months
  Efficacy will be evaluated by shortening of QRS duration on ECG.
Improvement of left ventricle ejection fraction | From enrollment to the end of follow-up period at 12 months
  Efficacy will be evaluated by increasing of left ventricle ejection fraction, measured by transthoracic echocardiography in 4 chamber apical position by Simpson's approach.
Decreasing of left ventricle end-diastolic diameter | From enrollment to the end of follow-up period at 12 months
  Efficacy will be evaluated by decreasing of left ventricle end-diastolic diameter measured by transthoracic echocardiography in parasternal long axis.
Decreasing of left ventricle end-diastolic volume | From enrollment to the end of follow-up period at 12 months
  Efficacy will be evaluated by decreasing of left ventricle end-diastolic volume measured by transthoracic echocardiography in apical 4-chamber position
Decreasing of left ventricle end-systolic volume | From enrollment to the end of follow-up period at 12 months
  Efficacy will be evaluated by decreasing of left ventricle end-systolic volume measured by transthoracic echocardiography in apical 4-chamber position
Improvement of mitral regurgitation | From enrollment to the end of follow-up period at 12 months
  Efficacy will be evaluated by decreasing of mitral regurgitation measured by transthoracic echocardiography in multiply positions

CONTACTS AND LOCATIONS:
Overall Officials: Yerlan Turubayev, MD, Principal Investigator — doctor
Locations (1):
- CF UMC, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tan JL, Lee JZ, Terrigno V, Saracco B, Saxena S, Krathen J, Hunter K, Cha YM, Russo AM. Outcomes of Left Bundle Branch Area Pacing for Cardiac Resynchronization Therapy: An Updated Systematic Review and Meta-analysis. CJC Open. 2021 Jun 16;3(10):1282-1293. doi: 10.1016/j.cjco.2021.05.019. eCollection 2021 Oct. PMID 34888508
- [Background] Goldenberg I, Kutyifa V, Klein HU, Cannom DS, Brown MW, Dan A, Daubert JP, Estes NA 3rd, Foster E, Greenberg H, Kautzner J, Klempfner R, Kuniss M, Merkely B, Pfeffer MA, Quesada A, Viskin S, McNitt S, Polonsky B, Ghanem A, Solomon SD, Wilber D, Zareba W, Moss AJ. Survival with cardiac-resynchronization therapy in mild heart failure. N Engl J Med. 2014 May 1;370(18):1694-701. doi: 10.1056/NEJMoa1401426. Epub 2014 Mar 30. PMID 24678999
- [Background] Yu CM, Lin H, Fung WH, Zhang Q, Kong SL, Sanderson JE. Comparison of acute changes in left ventricular volume, systolic and diastolic functions, and intraventricular synchronicity after biventricular and right ventricular pacing for heart failure. Am Heart J. 2003 May;145(5):E18. doi: 10.1016/S0002-8703(03)00071-1. PMID 12766742